CLINICAL TRIAL: NCT00421421
Title: A Randomised, Double-Blind, Placebo-Controlled, Multicentre Phase IV Study to Evaluate the Efficacy and Safety of Dutasteride 0.5mg Administered Orally Daily for 24 Weeks to Reduce The Risk of Acute Urinary Retention Relapse Following Successful Trial Without Catheter.
Brief Title: Effects Of Dutasteride On Risk Reduction Of Acute Urinary Retention Relapse Following Trial Without Catheter
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Incomplete information
Sponsor: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARI106807
Record Dates: First submitted 2007-01-11; First posted 2007-01-12 (Estimated); Last update posted 2007-11-27 (Estimated); Status verified 2007-11

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Acute Urinary Retention; Benign Prostatic Hyperplasia; Trial Without Catheter
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Dutasteride

INTERVENTIONS:
Drug: Dutasteride

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of dutasteride at reducing relapse rates of Acute Urinary Retention (AUR), including reduction in surgical intervention for benign prostatic hyperplasia (BPH), in patients who receive a 6 month treatment of dutasteride (0.5mg once daily) following a single episode of AUR followed by successful Trial Without Catheter compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Able to read, write and understand instructions related to study procedures and able to give written informed consent
* Able to swallow and retain oral medication
* Had a single, spontaneous episode of AUR related to BPH with a drained volume of between 500 and 1500ml
* Had a successful TWOC (defined as successful if the patient returns to satisfactory voiding within the first 24 hours after catheter removal without re-catheterisation) following 2 - 3 days treatment with alpha blocker (preferably alfuzosin 10mg OD) pre TWOC followed by up to seven days treatment with alpha blocker (preferably alfuzosin 10mg OD) post TWOC.
* Able to be randomised within 7 days of successful TWOC

Exclusion Criteria:

* Prostate volume (PV) of less than 30cc and greater than 80cc measured via Trans Rectal Ultrasound (TRUS) either at time of hospitalisation or as part of the screening / randomisation visit
* Previous episode of AUR prior to the current episode
* AUR not related to BPH i.e. postoperative retention following major abdominal / pelvis surgery
* Previous prostate or urethral surgery
* Previous positive prostate biopsy
* Any cause other than BPH that may result in urinary symptoms or changes in flow rates.
* Any unstable co-existing medical condition
* Previous 5-ARI use
* Previous alpha blocker treatment other than the study mandated 2 - 3 days pre and up to 7 days post TWOC period with alpha blocker (preferably alfuzosin 10mg OD)
* Use of prohibited meds (e.g. 5ARI's, anabolic steroids including testosterone, drugs with antiandrogenic properties)
* Liver enzymes (ALT, AST, ALP) at time of hospitalisation / screening visit greater than 2 x ULN or bilirubin at time of hospitalisation / screening visit greater than 1.5 x ULN.
* Serum creatinine at time of hospitalisation / screening visit greater than 1.5 x ULN
* Treatment with any other investigational product within 30 days prior to the first dose of study medication
* History or current evidence of alcohol or drug abuse within the last 12 months
* Prostate Specific Antigen (PSA) greater than 20ng/ml
* Use of suprapubic catheterisation after failed urethral catheterisation
* Neurogenic bladder dysfunction, confirmed or suspected, irrespective of etiology
* Isolated bladder neck disease
* Acute or chronic prostatitis
* Confirmed or suspected urethral stricture
* Known bladder stones
* Clot retention secondary to haematuria of any cause
* Patient unwilling to use a condom during sexual intercourse

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276
Dates: Start 2007-03

PRIMARY OUTCOMES:
Acute Urinary Retention (AUR) relapse rate during the 24 week treatment period | 24 Weeks

SECONDARY OUTCOMES:
Benign prostatic hyperplasia (BPH) related surgical intervention rates during study IPSS score during study Relationship between length of time of catheter in situ and Intravesical prostatic protrusion measurements on relapse rates | 24 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, BSc MBBS, Study Director — GlaxoSmithKline
Locations (25):
- United Kingdom (25):
  - GSK Clinical Trials Call Center, Barnet
  - GSK Clinical Trials Call Center, Bath
  - GSK Clinical Trials Call Centre, Birmingham
  - GSK Clinical Trials Call Center, Bradford
  - GSK Clinical Trials Call Center, Bristol
  - GSK Clinical Trials Call Center, Chester
  - GSK Clinical Trials Call Center, Colchester
  - GSK Clinical Trials Call Center, Crewe
  - GSK Clinical Trials Call Centre, Derby
  - GSK Clinical Trials Call Center, Edinburgh
  - GSK Clinical Trials Call Center, Glasgow
  - GSK Clinical Trials Call Center, Hull
  - GSK Clinical Trials Call Center, Leeds
  - GSK Clinical Trials Call Center, Leicester
  - GSK Clinical Trials Call Center, London
  - GSK Clinical Trials Call Center, Newcastle upon Tyne
  - GSK Clinical Trials Call Center, Nottingham
  - GSK Clinical Trials Call Center, Oldham
  - GSK Clinical Trials Call Center, Ormskirk
  - GSK Clinical Trials Call Center, Plymouth
  - GSK Clinical Trials Call Center, Stevenage
  - GSK Clinical Trials Call Center, Sunderland
  - GSK Clinical Trials Call Center, Sutton Coldfield
  - GSK Clinical Trials Call Center, Torquay
  - GSK Clinical Trials Call Center, Wakefield